CLINICAL TRIAL: NCT04936178
Title: A Multicenter Phase 1, Open-Label Study of NB003 to Assess Safety, Tolerability, Pharmacokinetics and Efficacy in Patients With Advanced Malignancies
Brief Title: A Study of NB003 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ningbo Newbay Technology Development Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB003-01
Record Dates: First submitted 2021-06-03; First posted 2021-06-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Phase and Dose Expansion Phase (Experimental): Dose escalation cohort:
  NB003 tablets will be administered orally twice daily for repeated 28-day cycles until discontinuation criteria are met.
  RP2D: one or more putative RP2D(s) will be explored in dose escalation phase with approximately 15 patients for each provisional RP2D(s)
  Dose expansion phase:
  In the dose expansion phase, additional patients will be enrolled at RP2D to further explore the safety, tolerability, PK, efficacy and biological activity of NB003 in specific disease cohorts, including GIST and other malignancies harboring genomic alterations of KIT or PDGFRα.
  Interventions: Drug: NB003 tablets

INTERVENTIONS:
Drug: NB003 tablets — NB003 tablets will be administered at assigned doses for escalation phase and RP2D doses for expansion phase orally twice daily for repeated 28-day cycles until discontinuation criteria are met.

SUMMARY:
This a A Phase 1, Open-label, Multicenter Study to Assess the Safety, Tolerability, and Pharmacokinetics of NB003 in Subjects with Advanced Malignancies

DETAILED DESCRIPTION:
This is a phase 1, open-label, multicenter study of NB003 which comprised of a dose escalation phase to determine the MTD or maximum administered dose (MAD), and the RP2D and a dose expansion phase to further explore the safety, PK and efficacy of NB003.

The dose escalation phase will enroll patients with advanced gastrointestinal stromal tumor (GIST) who have progressed on or had an intolerability to imatinib and other standard of cares (SoCs) or refused other SoCs, and patients with advanced malignancies other than GIST that harbors KIT or PDGFRα gene alterations who have relapsed or have refractory disease without an available effective therapy. The number of patients to be enrolled during the dose escalation part will vary depending on the underlining dose-toxicity curve and the number of dose levels tested prior to reaching MTD or MAD. After the MTD or MAD has been determined, based on emerging safety/PK data, one or more putative RP2D(s) will be explored in dose escalation phase with approximately 15 patients for each provisional RP2D(s) to establish the RP2D for dose expansion phase. This step will be regarded as RP2D confirmation part of dose escalation phase.

In the dose expansion phase, additional patients will be enrolled to further explore the safety, tolerability, PK, efficacy and biological activity of NB003 in specific disease cohorts, including GIST and other malignancies harboring genomic alterations of KIT or PDGFRα. Dose expansion phase is planned to investigate NB003 at the RP2D determined from dose escalation phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of any race ≥18 years age.
2. Histologically-confirmed diagnosis of unresectable, relapsed or metastatic GIST or other advanced malignancies.

   1. For dose escalation phase:

      * GIST patients must have progressed on or had an intolerability to imatinib and other SoCs or refused other SoCs.
      * Patients with an advanced solid tumor other than GIST must have relapsed or had refractory disease without an available effective therapy and harbor KIT or PDGFRα gene alterations (central laboratory confirmation is not required for screening).
   2. For dose expansion phase:

   Cohort 1: GIST patients with KIT or PDGFRα gene mutations, must have progressed on or been intolerant to at least imatinib, sunitinib, regorafenib and ripretinib (≥ fifth line therapy setting); Cohort 2a: GIST patients with KIT or PDGFRα gene mutations, must have progressed on or been intolerant to imatinib and sunitinib, and who have not received additional systemic therapy for advanced GIST (third line therapy setting); Cohort 2b: GIST patients with KIT or PDGFRα gene mutations, must have progressed on or been intolerant to imatinib, sunitinib and regorafenib, and who have not received additional systemic therapy for advanced GIST (forth line therapy setting); Cohort 3: GIST patients with KIT or PDGFRα gene mutations, must have progressed on or been intolerant to imatinib and have not received additional systemic therapy for advanced GIST (second line therapy setting); Cohort 4: GIST patients with PDGFRα exon 18 mutation and must have progressed on or been intolerant to avapritinib; in the countries/regions where avapritinib is not SoC, avapritinib-naïve patients can be enrolled; Cohort 5: Unresectable or metastatic melanoma patients with demonstrated evidence for KIT gene mutation and/or amplification, must have progressed on or been intolerant to SoCs; Cohort 6: Patients with other advanced malignancies other than GIST or melanoma which must be relapsed or refractory without an available effective therapy and harbor KIT or PDGFRα gene alterations.
3. For dose expansion phase: at least one measurable lesion per RECIST v1.1/mRECIST.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy ≥ 12 weeks.
6. Adequate organ and marrow function.
7. Tumor sample collection is required.

Exclusion Criteria:

1. Prior anti-cancer therapy within 2 weeks or at least 5 half-lives, whichever is longer, up to a maximum wash-out period of 21 days prior to the initiation of study drug administration.
2. Major surgery within 4 weeks of the first dose.
3. Radiotherapy with a limited field of radiation for palliation within 1 week prior to the first dose, with the exception as defined.
4. Patients currently receiving medications or herbal supplements known to be strong inhibitors or inducers of CYP3A4.
5. Patients currently receiving acid-reducing agents and are unable to stop use at least 2 weeks prior to the first dose.
6. Any known active central nervous system metastases and/or carcinomatous meningitis. Active infection including hepatitis B, hepatitis C, and HIV.
7. Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, uncontrolled pericardial effusion, uncontrolled pleural effusion, or any other conditions, which in the judgment of Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.
8. Any evidence of severe or uncontrolled systemic diseases which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | Approximately 24 months since the escalation first subject enrolled
  Dose Escalation Phase：Dose-limiting toxicities will be reviewed as a subset of adverse events that occur within the first 28 days of dosing and meet protocol-specified criteria.
Incidence of adverse events | Approximately 24 months since the escalation first subject enrolled; Approximately 26 months since the Expansion first subject enrolled
  Dose Escalation Phase and Dose Expansion Phase: An AE is any untoward medical occurrence in a participant who received study drug without regard to causal relationship.
Objective Response Rate (ORR) | Approximately 26 months since the Expansion first subject enrolled
  Dose Expansion Phase: Objective Response Rate (ORR) which is defined as the percentage of patients whose efficacy is confirmed as complete response(CR) or partial responses(PR)
Duration of Response(DOR) | Approximately 26 months since the Expansion first subject enrolled.
  Dose Expansion Phase: DOR is defined as the time from the date of first documented response until date of documented progression, for subjects who achieve CR or PR.

SECONDARY OUTCOMES:
Area under the curve (AUC) from time zero to the last measurable concentration AUC (0-t) | Approximately 24 months since the escalation first subject enrolled; Approximately 26 months since the Expansion first subject enrolled
  Dose Escalation Phase and Dose Expansion Phase: AUC (0-t) = Area under the serum concentration versus time curve from time zero (pre-dose) to the time of the last measurable concentration.
Maximum observed plasma concentration (Cmax) | Approximately 24 months since the escalation first subject enrolled; Approximately 26 months since the Expansion first subject enrolled
  Dose Escalation Phase and Dose Expansion Phase: Maximum observed plasma concentration (Cmax)
Time to Cmax (Tmax) | Approximately 24 months since the escalation first subject enrolled; Approximately 26 months since the Expansion first subject enrolled
  Dose Escalation Phase and Dose Expansion Phase: Time to Cmax (Tmax)
Terminal elimination half life | Approximately 24 months since the escalation first subject enrolled; Approximately 26 months since the Expansion first subject enrolled
  Dose Escalation Phase and Dose Expansion Phase: Terminal elimination half life
Objective Response Rate (ORR) | Approximately 24 months since the escalation first subject enrolled
  Dose Escalation Phase: Objective Response Rate (ORR) which is defined as the percentage of patients whose efficacy is confirmed as complete response(CR) or partial responses(PR)
Duration of Response(DOR) | Approximately 24 months since the escalation first subject enrolled
  Dose Escalation Phase: DOR is defined as the time from the date of first documented response until date of documented progression, for subjects who achieve CR or PR.

OTHER OUTCOMES:
Cancer relevant gene mutations | Approximately 24 months since the escalation first subject enrolled; Approximately 26 months since the Expansion first subject enrolled
  Dose Escalation Phase and Dose Expansion Phase:Cancer relevant gene mutations

CONTACTS AND LOCATIONS:
Locations (32):
- United States (6):
  - Standford University, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, Long Island City, New York
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - U T MD Anderson Cancer Center Investigational Pharmacy Services, Houston, Texas
- China (19):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guandong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guandong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Xiangya Hospital, Central South University, Changsha, Huanan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'An Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University school of medicine, Hangzhou, Zhejiang
- France (2):
  - Centre Léon Bérard, Lyon, Rhone
  - Institut Gustave Roussy, Villejuif, Val de Marne
- South Korea (2):
  - Asan Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid, Madrid
- Royal Marsden Hospital-London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No